CLINICAL TRIAL: NCT05736211
Title: Organization-level Youth Engagement Approach for Substance Misuse Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00091590; 5K01DA048201-03 (NIH)
Record Dates: First submitted 2023-02-09; First posted 2023-02-21 (Actual); Results first posted 2025-10-31 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2024-12

CONDITIONS: Drug Use; Substance Use; Opioid Use; Substance Misuse
Keywords: Adolescents; Young adults; Prevention; Youth Engagement; Randomized control trial
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): In this arm the study will implement an organization-level Youth Engagement prevention strategy by systematically incorporating Youth Engagement into prevention efforts in a community setting. Youth (individuals) participating in the intervention organizations' programming following the organization's completion of the YE intervention will complete surveys.
  Interventions: Behavioral: Organization-level Youth Engagement prevention strategy
- Control group (No Intervention): This arm will receive no intervention. Control group organizations will continue their normal prevention strategy without the inclusion of a Youth Engagement component

INTERVENTIONS:
Behavioral: Organization-level Youth Engagement prevention strategy — Systematically incorporating Youth Engagement into prevention efforts in a community setting
  Arms: Intervention group

SUMMARY:
This study will consist of a small pilot Randomized Controlled Trial (RCT). Four prevention organizations will be randomized either to include Youth Engagement in prevention efforts (treatment) or not (control). The study team will attempt to match the treatment and control groups on relevant characteristics such as geographic location (e.g., urban, rural), population served (e.g., church-based, school-based), and/or prior Youth Engagement involvement. The objective of this study is to evaluate the preliminary effectiveness of YE as a prevention strategy for opioid misuse in a small pilot randomized control trial (RCT). This pilot study will examine the effects of the YE prevention strategy on (a) organization-level outcomes, such as perceived value added to prevention programming and (b) individual-level outcomes such as personal skills and attitudes as well as knowledge and attitudes about substances including opioids. Up to 15 leaders/staff and 45 youth/young adults (60 people overall) will be recruited for the study.

DETAILED DESCRIPTION:
Substance misuse is a major public health problem and opioid misuse is an acute problem in rural and high poverty communities. Adolescence and young adulthood is a formative time for positive social development, as young people increase their needs for maturity and autonomy, define their identities, and carve out their roles in society. But many youth and young adults are isolated within communities, feel that they do not matter, and lack meaningful opportunities to engage with society and form positive connections with prosocial institutions. Further, community systems and settings that serve youth and young adults often do not effectively involve them. Engaging youth and young adults in their communities and in the prevention systems targeting substance misuse may prevent the use of substances by targeting two pathways. The first is an individual pathway via bolstering psychosocial development and reducing risks for opioids by providing youth and young adults with meaningful prosocial opportunities to fulfill developmental needs. The second is an environmental pathway via affecting health system and community-based settings through improving prevention efforts targeting young adults. This project tests an organization-level Youth Engagement (YE) approach to improve prevention.

Only organizations randomized to treatment will include youth/Young Adult (YA) participants. Youth/YA survey data will be collected at the start of their participation in the YE strategy (pre-YE) and 6 months later (post-YE). At the post-YE the study team will interview a subset of interested YE group participants to qualitatively assess their experiences and to identify, in their own voices, what aspects of YE emerge as important to youth development and their health-related decision-making.

The timeframe for this phase will be 12-18 months.

ELIGIBILITY:
INCLUSION CRITERIA:

Organizational leaders/staff:

* Leaders or staff of community-based prevention organizations based in North Carolina
* Organizations are youth/young adult-serving and focused on opioid misuse prevention
* Organizations demonstrate readiness, interest, need, and resources to invest in Youth Engagement as part of prevention
* Leaders or staff are or would be involved in implementing Youth Engagement strategy at the organization
* Leaders or staff are able to speak and read English fluently

Youth/young adult participants involved with organizations:

* Adolescents and young adults age 11 - 29
* Interested in participating in Youth Engagement with the community organization
* Able to speak and read English fluently

EXCLUSION CRITERIA:

• Organizations already incorporating a high level of Youth Engagement in its prevention work

Min Age: 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2024-03-14 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Parissa J Ballard, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest School of Medicine, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available. The information collected about organizations and from individual participants will be kept confidential; only aggregate results will be reported in manuscripts and reports.

REFERENCES:
- [Background] Erikson, E. H. Identity: Youth and crisis. (WW Norton & Company, 1968).
- [Background] Eccles JS, Midgley C, Wigfield A, Buchanan CM, Reuman D, Flanagan C, Iver DM. Development during adolescence. The impact of stage-environment fit on young adolescents' experiences in schools and in families. Am Psychol. 1993 Feb;48(2):90-101. doi: 10.1037//0003-066x.48.2.90. PMID 8442578
- [Background] Farrow JA. Youth alienation as an emerging pediatric health care issue. Am J Dis Child. 1991 May;145(5):491-2. doi: 10.1001/archpedi.1991.02160050015002. No abstract available. PMID 2042607
- [Result] Eccles, J. S. et al. Control versus autonomy during early adolescence. Journal of Social Issues 47, 53-68 (1991).

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Organization
Groups:
- Intervention Group: In this arm the study will implement an organization-level Youth Engagement prevention strategy by systematically incorporating Youth Engagement into prevention efforts in a community setting with 2 youth prevention organizations randomized to this arm. Participants will include organizational leaders/staff. Upon completion of the organization intervention. Youth (individuals) participating in the intervention organizations' programming will complete surveys.
- Control Group: This arm will receive no intervention. Organizations randomized to the control group will continue their normal prevention strategy without the inclusion of a Youth Engagement component. Participants will include organizational leaders/staff.
Period: Overall Study
Arm/Group | Intervention Group | Control Group
Started | 36; 2 Organization | 7; 2 Organization
Completed | 30; 2 Organization | 7; 2 Organization
Not Completed | 6; 0 Organization | 0; 0 Organization
Not completed — Lost to Follow-up | 6 | 0

BASELINE CHARACTERISTICS:
Groups:
- Intervention: In this arm the study will implement an organization-level Youth Engagement prevention strategy by systematically incorporating Youth Engagement into prevention efforts in a community setting.
  Organization-level Youth Engagement prevention strategy: Systematically incorporating Youth Engagement into prevention efforts in a community setting
- Control: This arm will receive no intervention. Control group organizations will continue their normal prevention strategy without the inclusion of a Youth Engagement component
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 36 | 7 | 43
Age, Customized [Count of Participants; unit: Participants]
  Age categories: 18 to 29 years | 2 | 2 | 4
  Age categories: 30 to 39 years | 3 | 1 | 4
  Age categories: 40 to 49 years | 1 | 1 | 2
  Age categories: 50 to 59 years | 0 | 1 | 1
  Age categories: 60 years or older | 0 | 2 | 2
  Age categories: 11 to 17 years | 30 | 0 | 30
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex: Female, Male: Female | 28 | 5 | 33
  Sex: Female, Male: Male | 7 | 2 | 9
  Sex: Female, Male: Missing data | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 12 | 0 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 0 | 7
  White | 9 | 5 | 14
  More than one race | 5 | 2 | 7
  Unknown or Not Reported | 3 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Staff Surveys--Youth Engagement (YE) Prevention Programming Value
Description: This outcome will be assessed through a survey measure administered to the organization leaders and staff in the YE intervention organizations only. The survey measures will be on a 1-5 scale with a higher score meaning a higher perceived programming value.
Time Frame: Month 6
Population: The population for this outcome is the YE intervention organizations only (intervention arm only).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 4
score on a scale | 4 (.816)

2. Primary Outcome: Perceived Retention of Youth/Young Adults in Youth Engagement (YE) Prevention Programming
Description: This outcome will be assessed through a survey measure on a 1-5 scale administered to the organization leaders and staff in the YE intervention organizations only, with higher scores indicated better retention.
Time Frame: Month 6
Population: The population for this outcome is the organization leaders and staff in the YE intervention organizations only (intervention arm only).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 4
score on a scale | 4.5 (.577)

3. Primary Outcome: Perceived Usefulness of Youth Engagement (YE) Prevention
Description: This outcome will be assessed through a survey measure administered to the organization leaders and staff in the YE intervention organizations only. The survey items will ask about perceived usefulness of the YE intervention for youth/young adults, the organization, and the community. Items will be on a 1-5 scale with higher scores indicating higher perceived usefulness.
Time Frame: Month 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 4
score on a scale
  Usefulness of YE intervention to youth/young adults | 4 (.816)
  Usefulness of YE intervention to organization | 4 (.816)
  Usefulness of YE intervention to community | 3.75 (.957)

4. Primary Outcome: Perceived Effectiveness, Quality, Reach, and Usefulness of General Prevention Approaches
Description: This outcome will be assessed through a survey measure administered to the organization leaders and staff in the Youth Engagement (YE) intervention organizations and comparison organizations. The survey measures will be on a 1-5 scale with higher scores indicating higher perceived quality, reach, and usefulness.
Time Frame: Month 6
Population: The population for this outcome is organization leaders and staff in both YE intervention and control organizations (intervention and control arms only).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 4 | 7
score on a scale
  Effectiveness of general prevention approaches | 3.50 (.577) | 3.71 (.951)
  Quality of general prevention approaches | 3.75 (.50) | 3.86 (1.07)
  Reach of general prevention approaches | 3.75 (.957) | 3.71 (1.1)
  Usefulness of general prevention approaches | 3.75 (.500) | 3.86 (1.22)

5. Secondary Outcome: Youth/Young Adults: Leadership and Communication Skills
Description: This outcome will be assessed through a survey measure administered to young adults involved in the youth engagement (YE) intervention at baseline (pre-YE) and 6 months later (post-YE). The survey measures will be on a 1-5 scale with higher scores indicating greater leadership and communication skills .
Time Frame: Baseline and Month 6
Population: The population for this outcome is the youth/young adult participants only (youth organizational participants arm).
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Youth Organizational Participants: Youth participating in the intervention organization's programming following the organization's completion of the YE intervention.
Arm/Group | Youth Organizational Participants
Number analyzed (Participants) | 26
score on a scale
  Youth Pre survey | 3.8 (.64)
  Youth Post survey | 4.0 (.55)

6. Secondary Outcome: Youth/Young Adults: Self-efficacy
Description: This outcome will be assessed through a survey measure administered to young adults involved in the youth engagement (YE) intervention at baseline (pre-YE) and 6 months later (post-YE). The survey measures will be on a 1-5 scale with higher scores indicating higher self-efficacy.
Time Frame: Baseline and Month 6
Population: The population for this outcome is the youth/young adult participants only (youth organizational participants arm).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Youth Organizational Participants
Number analyzed (Participants) | 26
score on a scale
  Youth pre-survey | 3.77 (.39)
  Youth post-survey | 4.10 (.45)

7. Secondary Outcome: Youth/Young Adults: Self Esteem
Description: This outcome will be assessed through a survey measure administered to young adults involved in the youth engagement (YE) intervention at baseline (pre-YE) and 6 months later (post-YE). The survey measures will be on a 1-5 scale with higher scores indicating greater self esteem.
Time Frame: Baseline and Month 6
Population: The population for this outcome is the youth/young adult participants only (youth organizational participants arm).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Youth Organizational Participants
Number analyzed (Participants) | 24
score on a scale
  Youth pre-survey | 3.30 (.58)
  Youth post-survey | 3.54 (.76)

8. Secondary Outcome: Youth/Young Adults: Social Connectedness
Description: This outcome will be assessed through a survey administered to young adults involved in the youth engagement YE intervention at baseline (pre-YE) and 6 months later (post-YE). The survey measures will be on a 1-5 scale with higher scores indicating greater social connectedness.
Time Frame: Baseline and Month 6
Population: The population for this outcome is the youth/young adult participants only (youth organizational participants arm).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Youth Organizational Participants
Number analyzed (Participants) | 26
score on a scale
  Youth pre-survey | 4.25 (.70)
  Youth post-survey | 4.26 (.62)

9. Secondary Outcome: Youth/Young Adults: Meaningful Social Role
Description: This outcome will be assessed through a survey measure administered to young adults involved in the youth engagement (YE) intervention at baseline (pre-YE) and 6 months later (post-YE). The survey measures will be on a 1-5 scale with higher scores indicating higher perceived meaningful social role.
Time Frame: Baseline and Month 6
Population: The population for this outcome is the youth/young adult participants only (youth organizational participants arm).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Youth Organizational Participants
Number analyzed (Participants) | 26
score on a scale
  Youth pre-survey | 4.03 (.54)
  Youth post-survey | 4.20 (.62)

10. Secondary Outcome: Youth/Young Adults: Beliefs and Intentions Related to Substance Use
Description: This outcome will be assessed through a survey measure administered to young adults involved in the youth engagement (YE) intervention at baseline (pre-YE) and 6 months later (post-YE). The survey measures will be on a 1-5 scale with higher scores indicating safer beliefs about perceived risks.
Time Frame: Baseline and Month 6
Population: The population for this outcome is the youth/young adult participants only (youth organizational participants arm).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Youth Organizational Participants
Number analyzed (Participants) | 25
score on a scale
  Youth pre-survey | 2.74 (.32)
  Youth post-survey | 2.75 (.37)

11. Other Pre Specified Outcome: Exploratory--Youth Engagement Prevention Programming Value, Qualitative
Description: This exploratory outcome will be assessed qualitatively through interviews with organizational leaders and staff
Time Frame: Month 6
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Exploratory--Retention of Youth/Young Adults in Youth Engagement Prevention Programming, Qualitative
Description: This exploratory outcome will be assessed qualitatively through interviews with organizational leaders and staff
Time Frame: Month 6
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Exploratory--Reach of Youth Engagement Prevention Efforts in the Community, Qualitative
Description: This exploratory outcome will be assessed qualitatively through interviews with organizational leaders and staff
Time Frame: Month 6
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Exploratory--Perceived Usefulness of Youth Engagement Prevention, Qualitative
Description: This exploratory outcome will be assessed qualitatively through interviews with organizational leaders and staff
Time Frame: Month 6
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Exploratory--Perceived Effectiveness, Quality, Reach, and Usefulness of General Prevention Approaches, Qualitative
Description: This exploratory outcome will be assessed qualitatively through interviews with organizational leaders and staff
Time Frame: Month 6
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Baseline through month 6
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/7
Other Adverse Events (participants affected / at risk) | 0/36 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-09-19): https://cdn.clinicaltrials.gov/large-docs/11/NCT05736211/Prot_SAP_000.pdf
  • Informed Consent Form (2025-06-17): https://cdn.clinicaltrials.gov/large-docs/11/NCT05736211/ICF_001.pdf